CLINICAL TRIAL: NCT05323903
Title: The Effect of Game-Based Learning and Telesimulation Application on Nursing Students' Self-Efficacy in Knowledge, Skills, Motivation and Clinical Performance in Postpartum Hemorrhage Management
Brief Title: The Effect of Game-Based Learning and Telesimulation on Nursing Students' Management of Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Yesim CETINKAYA SEN, Principal Investigator, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-109
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): Postpartum Hemorrhage and Its Management course
- Intervention Group 1- Telesimulation (Experimental): Postpartum Hemorrhage and Its Management course, Telesimulation application
  Interventions: Other: Telesimulation
- Intervention Group 2- Kahoot (Experimental): Postpartum Hemorrhage and Its Management course, Kahoot game
  Interventions: Other: Kahoot Game
- Intervention Group 3-Telesimulation and Kahoot (Experimental): Postpartum Hemorrhage and Its Management course, Telesimulation application and Kahoot game
  Interventions: Other: Telesimulation; Other: Kahoot Game

INTERVENTIONS:
Other: Telesimulation — Telesimulation is an application that is a teaching process by which telecommunication and healthcare simulation resources are used to provide education, training and assessment to learners at an off-site location. In this study, simulation was recorded and this was shared with the students through means of telecommunication.
  Arms: Intervention Group 1- Telesimulation; Intervention Group 3-Telesimulation and Kahoot
Other: Kahoot Game — Kahoot is a game-based learning platform, used as educational technology in schools and other educational institutions.
  Arms: Intervention Group 2- Kahoot; Intervention Group 3-Telesimulation and Kahoot

SUMMARY:
This study was conducted to evaluate the effects of Kahoot and telesimulation methods on the knowledge, skills, motivation and clinical performance of nursing students in the management of postpartum hemorrhage and to examine the students' views on these methods.

This is a randomized controlled intervention study in which the quantitative research method is used. The study sample consisted of year-2 students (n=177) who took the Obstetrics and Gynecology Nursing course in the spring semester of the 2020-2021 academic year at the Faculty of Gulhane Nursing at SBU. The control group consisted of 44 students, and the intervention group was divided into three groups and randomized to include 44 students in each group, with a total of 133 students. All students attended the "Postpartum Hemorrhage and its Management" course, and after the course, Group II received the telesimulation intervention, Group III the Kahoot game intervention and Kahoot game and telesimulation to Group IV. The control group did not receive any intervention.

DETAILED DESCRIPTION:
This study was conducted to evaluate the effects of Kahoot and telesimulation methods on the knowledge, skills, motivation and clinical performance of nursing students in the management of postpartum hemorrhage and to examine the students' views on these methods.

This is a randomized controlled intervention study in which the quantitative research method is used. The study sample consisted of year-2 students (n=177) who took the Obstetrics and Gynecology Nursing course in the spring semester of the 2020-2021 academic year at the Faculty of Gulhane Nursing at SBU. The control group consisted of 44 students, and the intervention group was divided into three groups and randomized to include 44 students in each group, with a total of 133 students. All students attended the "Postpartum Hemorrhage and its Management" course, and after the course, Group II received the telesimulation intervention, Group III the Kahoot game intervention and Kahoot game and telesimulation to Group IV. The control group did not receive any intervention.

All the practices were carried out remotely with students who had their education through distance learning due to COVID-19. Groups were formed from the students according to randomization. The student names whose groups were determined were assigned to their own group in Microsoft Teams. The application phase of the study included the pre-test, theoretical education on Postpartum Hemorrhage, playing games on the Kahoot platform, telesimulation application, and post-test application to all groups.

The "Postpartum Hemorrhage and its Management" course was held on March 9, 2021, in two 40-minute sessions, using PowerPoint as training material, synchronized with the whole class over Microsoft Teams. After all the content for the Kahoot game was prepared, the students were briefed through a synchronous 30-minute online meeting in Microsoft Teams with a PowerPoint presentation on how to log in to Kahoot and how to play the games. An entry guide to Kahoot has been prepared and distributed to the students. Then, on April 26, 2021, five different Kahoot games for Group 3 and Group 4 were uploaded and a PIN was sent to the students to play one game per day. After the Kahoot game was over, Telesimulation Application was carried out with Group 2 and Group 4. After the telesimulation application, the final tests were conducted.

ELIGIBILITY:
Inclusion Criteria:

* Taking the Obstetrics and Gynecology Nursing Course for the first time,
* Having no professional experience,
* Having a smartphone, tablet or computer with an internet connection,
* Continuing the course with distance learning during the COVID-19 pandemic period,
* Receiving education on Postpartum Hemorrhage for the first time,
* Voluntarily accepting to participate in the study.

Exclusion Criteria:

* Not attending the theoretical lesson,
* Not playing the game that was sent to them,
* Not volunteering to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Instructional Materials Motivation Survey | 2 Months
  The Instructional Materials Motivation Survey (IMMS) aims to assess the motivational characteristics of instructional materials or courses using the Attention, Relevance, Confidence, and Satisfaction (ARCS) model of motivation. It was developed by Keller et al. in 2006. The five-point Likert type scale consists of 36 items in the original scale. In the last Turkish adaptation study by Dinçer and Doğanay, 3 of the items were excluded from the original scale and a total of 33 items were included in the Turkish version of the scale.
Self-Efficacy in Clinical Performance Scale | 2 Months
  The scale, developed by Cheraghi et al. in 2009, is used to measure the self-efficacy of the nurses in order to predict their clinical performance. It is a Likert type scale with 37 items in total under 4 factors, which are assessment, diagnosis and planning, implementation, and evaluation.

SECONDARY OUTCOMES:
Postpartum Hemorrhage Telesimulation Skill Evaluation Form | 2 Months
  The form, developed by the researcher in line with the literature, consists of a total of 30 items under 6 sub-dimensions. These are as follows: Patient admission and evaluation(3 items), communication(3 items), physical examination(3 items), signs and symptoms of hypovolemic shock(6 items), postpartum hemorrhage protocol(13 items) and blood transfusion(2 items). If the student stated the expected practical steps in postpartum hemorrhage, it is scored 1, if not, 0 points are given. In the form, the lowest score is "0" and the highest score is "30" (min=0, max=30).

CONTACTS AND LOCATIONS:
Overall Officials: Gülten GÜVENÇ, Prof., Study Director — Department of Obstetrics and Gynecology Nursing, Gulhane Nursing Faculty, Health Sciences University
Locations (1):
- Istanbul Sağlık Bilimleri Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No